CLINICAL TRIAL: NCT01051986
Title: A Randomized Comparison of the SAphenous VEin Versus Right Internal Thoracic Artery as a Y-Composite Graft (SAVE-RITA Trial)
Brief Title: A Prospective Randomized Study for Comparison of Y-Composite Grafts
Acronym: SAVERITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ki-Bong Kim, Professor and Chairman, Department of Thoracic and Cardiovascular Surgery, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-0803-024-237
Record Dates: First submitted 2010-01-17; First posted 2010-01-20 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass; off-pump surgery; composite graft; saphenous vein; internal thoracic artery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SVG group (Active Comparator): patients who underwent off-pump coronary artery bypass using saphenous vein composite grafting based on the left internal thoracic artery
  use saphenous vein as a composite graft connected to the left internal thoracic artery
  Interventions: Procedure: saphenous vein composite grafting
- RITA group (Active Comparator): patient who underwent off-pump coronary artery bypass using right internal thoracic artery composite grafting based on the left internal thoracic artery
  use right internal thoracic artery as a composite graft connected to the left internal thoracic artery
  Interventions: Procedure: right internal thoracic artery composite grafting

INTERVENTIONS:
Procedure: saphenous vein composite grafting — use saphenous vein as a composite graft connected to the left internal thoracic artery
  Other Names: SAVERITA SVG
  Arms: SVG group
Procedure: right internal thoracic artery composite grafting — right internal thoracic artery is used as a composite graft connected to the left internal thoracic artery
  Other Names: SAVERITA RITA
  Arms: RITA group

SUMMARY:
The purpose of this study is to compare early and 1-year graft patency rates of saphenous vein composite grafts with those of right internal thoracic artery composite graft and mid-term clinical outcomes in patients who undergo off-pump coronary artery bypass grafting(OPCAB). We also evaluate microscopic findings of saphenous vein graft harvested no touch technique and used as composite graft.

DETAILED DESCRIPTION:
The SAVERITA trial was designed as a randomized, controlled trial to recruit 224 patients who undergo off-pump coronary artery bypass using Y-composite graft based on the left internal thoracic artery. Patients were randomized by use of a randomization table. Composite conduit was made using saphenous vein or right internal thoracic artery according to the randomization result. The primary end point is to evaluate early and 1-year postoperative graft patency. The secondary end points are overall survival, freedom from cardiac death and freedom from MACCE(major adverse cardiac or cerebrovascular events). In saphenous vein group, 20 remnant saphenous vein specimen was evaluated histologically to compare the difference between composite grafted vein and manually dilated saphenous vein.

ELIGIBILITY:
Inclusion Criteria:

* age equal or more than 40
* age equal or less than 75
* patients who agree to the enrollment

Exclusion Criteria:

* Patients with heart failure (left ventricular ejection fraction < 25%)
* patients who have intractable ventricular arrhythmia
* patients who has been treated for cancer
* patients who has infectious disease
* patients who are planned to undergo combined cardiac surgery
* patients who has medical co-morbidity with expected survival less than 1 year
* patients who has a problem using right internal thoracic artery or saphenous vein
* patients with a history of previous cardiac surgery
* Patients with chronic renal failure
* patients who undergo emergency operation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Bong Kim, MD, PhD, Principal Investigator — Department of throacic and cardiovascular surgery, Seoul National University Hospital
Locations (1):
- Seoul National Uinversity Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim KB, Hwang HY, Hahn S, Kim JS, Oh SJ. A randomized comparison of the Saphenous Vein Versus Right Internal Thoracic Artery as a Y-Composite Graft (SAVE RITA) trial: One-year angiographic results and mid-term clinical outcomes. J Thorac Cardiovasc Surg. 2014 Sep;148(3):901-7; discussion 907-8. doi: 10.1016/j.jtcvs.2014.03.057. Epub 2014 May 16. PMID 24973924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients, 40 to 75 years of age, who were scheduled to between September 2008 and October 2011 patients who undergo off-pump CABG (OPCAB) for multivessel coronary artery disease using a Y-composite graft based on the in situ left ITA were evaluated for eligibility
Pre-assignment Details: Exclusion criteria included patients with ineligible Y-composite graft revascularization, unavailable RITA or SV, left ventricular dysfunction, chronic renal failure requiring renal replacement therapy, a history of previous cardiac operation, emergency, or a medical history that might limit the possibility of mid-term follow-up
Groups:
- RITA Group: patient who underwent off-pump coronary artery bypass using right internal thoracic artery composite graft based on the left internal thoracic artery
  use right internal thoracic artery as a composite graft connected to the left internal thoracic artery
  right internal thoracic artery composite grafting : right internal thoracic artery is used as a composite graft connected to the left internal thoracic artery
- SVG Group: patients who underwent off-pump coronary artery bypass using saphenous vein composite graft based on the left internal thoracic artery
  use saphenous vein as a composite graft connected to the left internal thoracic artery
  saphenous vein composite grafting : use saphenous vein as a composite graft connected to the left internal thoracic artery
Period: Overall Study
Arm/Group | RITA Group | SVG Group
Started | 112 | 112
Completed | 107 | 108
Not Completed | 5 | 4
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RITA Group | SVG Group | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 58 | 121
  >=65 years | 49 | 54 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.0) | 63.3 (7.8) | 63.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 30 | 51
  Male | 91 | 82 | 173
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 112 | 112 | 224

OUTCOME MEASURES:

1. Primary Outcome: 1 Year Graft Patency Rates
Description: 1 year graft patency of second limb conduits measured by 1 year coronary angiography
Time Frame: one year
Measure: Number; unit: percentage of distal anastomoses
Units Other Than Participants: distal anastomosis
Arm/Group | RITA Group | SVG Group
Number analyzed (Participants) | 107 | 108
Number analyzed (distal anastomosis) | 204 | 245
percentage of distal anastomoses | 97.1 | 97.1

2. Secondary Outcome: Overall Survival
Description: Overall survival rate at 4 years
Time Frame: 4 years
Measure: Number; unit: percentage of participiciants
Arm/Group | RITA Group | SVG Group
Number analyzed (Participants) | 112 | 112
percentage of participiciants | 97.8 | 97.6

3. Secondary Outcome: Freedom From Cardiac Death
Description: Freedom rate from cardiac death at 4 years
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | RITA Group | SVG Group
Number analyzed (Participants) | 112 | 112
percentage of participants | 100 | 99.1

4. Secondary Outcome: Freedom From MACCE(Major Adverse Cardiac and Cerebrovascular Events)
Description: freedom from MACCE(major adverse cardiac and cerebrovascular events)at 4 years
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Arm/Group | RITA Group | SVG Group
Number analyzed (Participants) | 112 | 112
percentage of participants | 91.1 | 94.4

5. Secondary Outcome: Early Angiographic Patency Rates
Description: The patency rate of the SV side-arm composite graft evaluated with coronary angiograms early after CABG
Time Frame: 1.4days
Measure: Number; unit: percentage of distal anastomoses
Units Other Than Participants: number of distal anastomoses
Arm/Group | RITA Group | SVG Group
Number analyzed (Participants) | 110 | 109
Number analyzed (number of distal anastomoses) | 208 | 248
percentage of distal anastomoses | 99.5 | 98.8

ADVERSE EVENTS:
Arm/Group | RITA Group | SVG Group
Serious Adverse Events (participants affected / at risk) | 8/112 | 6/112
Other Adverse Events (participants affected / at risk) | 0/112 | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RITA Group (N=112) | SVG Group (N=112)
Early death (Cardiac disorders) | 1 (1) | 0 (0) — death after surgery during the same hospital stay
Recurrent angina (Cardiac disorders) | 8 (8) | 4 (4) — angina recurrence during the follow up
Reintervefntion (Cardiac disorders) | 4 (4) | 1 (1)
Late death (Cardiac disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
the current study is not a multicenter "all-comers" study, although it is a prospective, randomized, controlled trial.

The 1-year graft patency rates and clinical outcomes of 34 months do not provide sufficient data to reach a definite conclusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No